CLINICAL TRIAL: NCT06023940
Title: Variability in Microbial Response to Dietary Fiber
Acronym: TRIUMPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Elizabeth Jane Parks, Professor, Nutrition & Exercise Physiology-MED, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2053546
Record Dates: First submitted 2023-05-04; First posted 2023-09-05 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Microbial Colonization
Keywords: colonoscopy; fiber
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Treatment group: 2 week high fiber diet Control group: no diet provided, subjects eat whatever they want
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Fiber (Experimental): Subjects are provided a high-fiber diet for 2 weeks. Tests include: blood biochemistries, body composition measured via DEXA, fecal sample collection, and anthropometrics measured
  Interventions: Dietary Supplement: High fiber
- Control (No Intervention): Subjects are not provided any diet, instead they eat what they choose for two weeks while they participate in a series of tests including: fecal sampling, food records, questionnaires/surveys, and anthropometrics

INTERVENTIONS:
Dietary Supplement: High fiber — A pea fiber supplement is added to a diet of regular foods. Participants receive 25g fiber daily.
  Arms: High Fiber

SUMMARY:
The goal of this clinical trial is to understand varying in responses to different dietary patterns in healthy people who are getting a health screening colonoscopy.

The main questions it aims to answer are:

* What is the variability in the change of the microbes in the gut of (1) a provided diet that is high in fiber vs (2) a diet of the participant's choice.
* What is the magnitude of fasting changes in glucose and lipids following the short-term, high-fiber feeding period and identify candidate predictive factors (short-chain fatty acids, BMI, sex, starting glucose level) for these changes

Participants will be in one of two groups:

1. High-fiber diet group: These participants will have a series of measurements that include: blood biochemistries, body composition measured via DEXA, anthropometrics, surveys and questionnaires, and collection of fecal samples.
2. Normal diet group: These participants will eat a diet that is of their choosing (ad libitum) and will have a series of measurements that include: fecal samples, and questionnaires/surveys including food records.

DETAILED DESCRIPTION:
Fiber fermentation in the colon produces short chain fatty acids (SCFA) and alters the microbial composition and activity. These effects may be mechanisms linking a high-fiber diet to improved health. However, different people may respond to dietary fiber differently and the variability in early, dietary-induced SCFA concentration changes has not been established. This lack of basic understanding in individual patterns of microbial SCFA production significantly limits efforts in the field of Precision Nutrition designed to target dietary strategies to improve health and advance lifestyle treatments in healthcare in the future. In this project, the central hypothesis is that the mechanisms by which dietary fiber provide metabolic benefits include a direct physical effect to improve fasting glucose and lipids and an effect related to increasing SCFA concentration. These are the ideas being tested in this study.

Using fiber derived from peas in a two-week human feeding intervention, Aim 1 will quantitate the variability in high-fiber-induced change in microbial composition and SCFA production by specifically testing the hypothesis that Following successful colonoscopy bowel prep, variability in the reduction in microbial species will be very small, while repopulation after a standardized high-fiber diet will be characterized by larger differences between individuals with regard to the quantity of bifidobacterial and the Firmicutes/ Bacteroidetes ratio.

Aim 2 will quantitate the magnitude of fasting changes in glucose and lipids following the short-term, high-fiber feeding period and identify candidate predictive factors (SCFA, BMI, sex, starting glucose level) for these changes by testing the hypothesis that a two-week, high-fiber diet will result in lower plasma glycemia and triglycerides. Participants (n=30) who have undergone a health-screening colonoscopy (HSC) are fed a high-fiber diet for 14 days. Fecal samples are collected before the colonoscopy and on days 1, 7 and 14 after the colonoscopy during high-fiber feeding. On day 1 and 14, the subject visits the clinical unit for a fasting blood draw (for measurement of glucose, lipids, and plasma SCFA), surveys and questionnaires.

A control arm will also be included as part of this study. The purpose of the control arm is to quantitate the variability in microbial composition and SCFA production from an ad libitum diet of participants. Instead of providing a high-fiber diet, the repopulation of the gut microbiome will be observed when participants eat a diet that is of their choosing. A series of food records and fecal samples pre- and post-procedure will be collected. Figure 2 shows the protocol of this arm. Food records will be collected: pre-procedure, days 0 (procedure day), 1, 2, 4, 7, 10, 13. Fecal collection will be collected: pre-procedure, 3, 5, 8, 11, 14. This arm will not include the blood collection or DEXA scan.

ELIGIBILITY:
Intervention Arm

Inclusion Criteria:

* Men and women
* Age 45-65y: the average age of people referred for a screening colonoscopy
* BMI ≥20.0 or ≤40.0 kg/m2
* Weight stable: no fluctuations in body weight of greater than 4 kg in the last 3 months
* Scheduled for a health-screening colonoscopy
* Willingness to consume a high-fiber diet
* Willing to provide blood and fecal samples
* Healthy or have one or more characteristics of the metabolic syndrome (but not diabetic) Metabolic syndrome criteria

  1. A large waistline: 35 inches or more for women 40 inches or more for men
  2. High triglycerides: 150 mg/dL or higher
  3. Low HDLc level: <50 mg/dL for women <40 mg/dL for men
  4. High blood pressure ≥130/85 mmHg
  5. Fasting blood sugar ≥100 mg/dL - Pre-diabetes acceptable (glucose <125 mg/dL or HbA1c <6.5%)
* Subjects are also eligible if they are stably treated with statin drugs, anti-hypertensive medications, and anti-depressants. These are eligible as long as the drug category does not alter appetite, body weight, or the microbiome (if known).

Exclusion Criteria:

* Pregnant or lactating, or planning to become pregnant
* BMI of <20.0 or >40.0 kg/m2
* Use of tobacco products
* Uncontrolled hypertension and blood pressure ≥ 180/110
* Use of medications that affect the gut microbiome (e.g., antibiotics)
* Taking medications known to affect appetite (phentermine) or gastrointestinal function (e.g. metformin)
* On a special diet vegetarian, or other restricted dietary patterns
* Undergoing weight loss
* Ad libitum intake of fiber above 25 g/day (mean intake in the US population is 17 g/day) and also an intake of fiber <10 g/d
* Ad libitum alcohol intake of greater than 7 drinks/week for women and 14 drinks/week for men
* History of disease (example colon cancer, etc.)
* Live more than 45 miles away from the University because participants will need to come into the Lab every 3 days or so to pick up meals.

Control Arm Inclusion criteria

* Men and women
* Age 45-65y: the average age of people referred for a screening colonoscopy
* Scheduled for a health-screening colonoscopy
* Willing to provide fecal samples
* Subjects are also eligible if they are stably treated with statin drugs, anti-hypertensive medications, and anti-depressants. These are eligible as long as the drug category does not alter appetite, body weight, or the microbiome (if known).

Exclusion criteria

* Pregnant or lactating, or planning to become pregnant
* Use of medications that affect the gut microbiome (e.g., antibiotics within the past 30 days)
* History of disease (example colon cancer, active GI bleeding, inflammatory bowel disease, etc.)
* Live more than 45 miles away from the University because participants will need to come into the Lab every 3 days or so to deliver fecal samples.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Variability in microbial composition as measured by 'alpha diversity' | 2 weeks
  Measured via fecal sample. Intervention group - measured once before scheduled health screening colonoscopy and 2 times over 2 weeks post-colonoscopy (day 1, 7, 14).
  Control group - measured once before scheduled health screening colonoscopy and 5 days over 2 weeks post-colonoscopy (day 3, 5, 8, 11, 14).
  Variability in microbial composition refers to how many different kinds of microbes are present in the fecal sample. We are testing the possibility that the more kinds of microbes, the healthier the person. The higher the measure the alpha diversity, the greater the number of different microbes.
Concentration of SCFA | 2 weeks
  Measured via fecal sample. Intervention group - measured once before scheduled health screening colonoscopy and 2 times over 2 weeks post-colonoscopy (day 1, 7, 14).
  Control group - measured once before scheduled health screening colonoscopy and 5 days over 2 weeks post-colonoscopy (day 3, 5, 8, 11, 14).

SECONDARY OUTCOMES:
Blood glucose concentration (mg/dL) | 2 weeks
  Measure changes in fasting blood glucose concentration following the short-term, high-fiber feeding period. Blood taken at screening, baseline, and follow up.
Blood lipid concentation (total cholesterol, LDLc, HDLc) (mg/dL) | 2 weeks
  Measure changes in fasting blood lipid concentration (mg/dL) following the short-term, high-fiber feeding period. Blood taken at screening, baseline, and follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Parks, Principal Investigator — University of Missouri-Columbia; Yezaz Ghouri, MD, Principal Investigator — University of Missouri-Columbia; Katherene Anguah, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No